CLINICAL TRIAL: NCT04452175
Title: Cigarette Consumption After switchinG to High or Low Nicotine strENght E-cigaretteS In Smokers With Schizophrenia Spectrum Disorders: A 12-month Randomised, Double-blind Multicentre Trial
Brief Title: Cigarette Consumption After switchinG to High or Low Nicotine strENght E-cigaretteS In Smokers With Schizophrenia
Acronym: GENESIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Collaborators: Juul Labs, Inc. (Industry); St. Petersburg State Pavlov Medical University (Other); Bashkir State Medical University (Other); Ukrainian Institute on Public Health Policy (Other); University of Surrey (Other); Eclat Srl. (Other)
Responsible Party: Principal Investigator, PASQUALE CAPONNETTO, Principal Investigator, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GENESIS, RCT UKRIT
Record Dates: First submitted 2020-06-24; First posted 2020-06-30 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Smoking; Schizophrenia Spectrum and Other Psychotic Disorders
MeSH Terms: conditions — Smoking; Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIGH 5% (Experimental)
  Interventions: Other: JUUL E-CIGARETTE
- LOW 1.7% (Active Comparator)
  Interventions: Other: JUUL E-CIGARETTE

INTERVENTIONS:
Other: JUUL E-CIGARETTE — JUUL E-CIGARETTE USAGE FOR 24 WEEKS

SUMMARY:
Smokers with schizophrenia spectrum disorders have high rates of morbidity and mortality from smoking-related diseases compared with the general population and current options for smoking cessation in this vulnerable group are unsatisfactory.

Considering that most people with schizophrenia spectrum disorders continue smoking, it is urgent to consider alternative and more efficient interventions to reduce or prevent their morbidity and mortality. Switching to combustion-free technologies for nicotine delivery (I.e. e-cigarettes) could be a pragmatic and much less harmful alternative to tobacco smoking with the possibility of significant health gains. Emerging research is suggesting that ECs may be useful for smoking cessation and relapse prevention in people with schizophrenia spectrum disorders. In particular, a study conducted with JUUL e-cigarette with 5% nicotine strength showed that this product had sufficient nicotine delivery and product appeal to determine high success rates in heavy smokers with schizophrenia spectrum disorders.

In consideration of these preliminary findings, we hypothesized that switching smokers with a schizophrenia spectrum disorder diagnosis to JUUL e-cigarette with 5% nicotine strength could result in higher success rates compared to JUUL e-cigarette with 1.7% nicotine strength. Recent work indicates that nicotine PK of the JUUL e-cigarette with 5% nicotine strength (a device that utilizes a nicotine salt formulation) approximates the nicotine delivery of combustible cigarettes and that the 5% nicotine strength product is far more efficient in delivering nicotine compared to the sister product with 1.7% nicotine strength. Both products are identical in their appearance, making them suitable for a double-blind study design.

DETAILED DESCRIPTION:
Multicenter, 12-months prospective trial, utilizing a randomized, double-blind, 2-arm parallel, switching design to compare effectiveness, tolerability, acceptability, and pattern of use between high (JUUL 5% nicotine) and low nicotine strength devices (JUUL 1.7% nicotine) in adult smokers with schizophrenia spectrum disorders. The study will take place at 5 international sites: UK (London), Italy (Catania), Russia (Ufa and St. Petersburg) and Ukraine (Kiev).

The two devices have identical appearance and will be assigned in a double-blind fashion. Study products will be provided for a total of 6-months (intervention phase); the intervention phase will be followed by a further 6-months observational period (follow-up phase) during which no products will be dispensed to participants. Throughout the follow-up phase and up to the final visit at 12-months, changes in smoking/vaping behavior and in their pattern of use will be tracked under naturalistic condition and compared between study groups. Any changes in symptom severity related to schizophrenia spectrum disorders within and between both arms of the study will be monitored. The intervention phase of the study will consist of a total of nine visits (including screening). The follow-up phase will consist of three additional visits (two telephone contacts and one final face to face visit).

In summary, the main objectives of the study will be to:

1. Quantify the proportion of continuous quitters among participants at 6-months in both arms of the study;
2. Quantify the proportion of continuous reducers among participants at 6-months in both arms of the study;
3. Quantify the proportion of continuous quitters among participants at 12-months in both arms of the study;
4. Quantify the proportion of continuous reducers among participants at 12-months in both arms of the study;
5. Compare continuous quit and reduction rates between study arms at 6- and 12-months;
6. Quantify adverse events throughout the whole duration of the interventional phase of the study in both arms;
7. Compare adverse events between study arms.

Additional objectives of the study will be to:

1. Measure Subjective perceptions and experiences of the two nicotine strenghts by the psychometrically validated modified Cigarette Evaluation Questionnaire - mCEQ (at 6-months);
2. Compare level of mCEQ between study arms (at 6-months);
3. Assess pattern of products use among participants throughout the whole duration of the study (both at intervention + follow-up phases) in both arms of the study;
4. Compare pattern of product use between study arms (both at intervention + follow-up phases).
5. Compare changes in symptom severity of patients with schizophrenia by Positive and Negative Syndrome Scale (PANSS) within and between both arms of the study (both at 6- and 12-months);
6. Compare changes in exercise tolerance by Chester Step Test within and between both arms of the study (only at 6-months);
7. Compare changes in weight/BMI within and between both arms of the study (both at 6- and 12-months);
8. Quantify self-rated mental health (SRMH) throughout the whole duration of the study (by means of a specifically designed APP) within and between both arms of the study (both at 6- and 12-months).

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18yrs)
* Regular smoking (>10 cigarettes a day; for at least one year)
* Exhaled breath CO (eCO) level > 7 ppm
* Not currently attempting to quit smoking or wishing to do so in the next 30 days; this will be verified at screening by the answer ''NO'' to the question ''Do you intend to quit in the next 30 days?''
* Schizophrenia spectrum disorder diagnosis (schizophrenia, delusional disorder, schizoaffective disorder, personality disorder, schizoid personality disorder, etc) by DSM-V criteria
* Understand and provide informed consent
* Able to comply with all study procedures

Exclusion Criteria:

* Institutionalized patients
* Acute decompensation of Schizophrenia spectrum disorder symptoms within the past month
* Change in antipsychotic treatment within the past month
* No recent history of hospitalization for any serious medical condition within 3 months prior to screening, as determined by the investigator.
* Myocardial infarction or angina pectoris within 3 months prior to screening, as determined by the investigator.
* Current poorly controlled asthma or COPD
* Pregnancy, planned pregnancy or breastfeeding. Any female participant who becomes pregnant during this study will be withdrawn.
* Participants who have a significant history of alcoholism or drug/chemical abuse within 12 months prior to screening, as determined by the investigator.
* Accepting to take part in a smoking cessation program
* Participants who regularly use any recreational nicotine (e.g. e-cigarettes,) or tobacco product (e.g. tobacco heated products, oral smokeless) other than their own cigarettes within 30 days of screening.
* Participants who have used smoking cessation therapies (e.g varenecline, buproprion, or NRT) within 30 days of screening.
* Participants who are still participating in another clinical study (e.g. attending follow-up visits) or who have recently participated in a clinical study involving administration of an investigational drug (new chemical entity) within the past 3 months.
* Participants who have, or who have a history of, any clinically-significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological or other major disorder that, in the opinion of the investigator or their appropriately qualified designee, would jeopardise the safety of the participant or impact on the validity of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-10-30 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Rates of participants with continuous smoking abstinence at 6-month | 24 WEEK
  self-reported continuous smoking abstinence at 6-month from the previous visit, biochemically verified by exhaled CO measurements of ≤ 7 ppm

SECONDARY OUTCOMES:
Rates of participants with continuous smoking abstinence at 12-month | 52 WEEK
Rates of participants with continuous smoking reduction at 6-month | 24 WEEK
Rates of participants with continuous smoking reduction at 12-month | 52 WEEK
Proportion of AEs | 24 WEEK
Absolute change in PANSS | 24 WEEK
Absolute change in mCEQ | 24 WEEK
Absolute change in Chester Step Test-derived values | 24 WEEK
Change in App-derived endpoints (self-rated mental health -SRMH). | 24 WEEK

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Caponnetto, Principal Investigator — University of Catania
Locations (1):
- CPCT, Catania, Italy